CLINICAL TRIAL: NCT06437821
Title: Comparative Effect of Graston Technique and Petrissage Technique on Tight Trapezius Muscles in Young Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/717
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Trapezius Muscle Strain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Petrissage (Other)
  Interventions: Diagnostic Test: Petrissage
- Graston Technique (Experimental)
  Interventions: Other: Graston Technique

INTERVENTIONS:
Diagnostic Test: Petrissage — The calf muscles will receive a firm, deep-circulation massage with fingertip pressure
  Arms: Petrissage
Other: Graston Technique — The calf muscles will receive a firm, deep-circulation massage with fingertip pressure
  Arms: Graston Technique

SUMMARY:
This research aims to contribute valuable insights into the potential benefits of incorporating the portable wedge device into preventive or therapeutic interventions for calf-related musculoskeletal issues. By combining economical, ergonomic principles and user-friendly features, the proposed device offers individuals a convenient and efficient means to enhance their calf flexibility, ultimately mitigating strain and reducing spasms.

DETAILED DESCRIPTION:
Developing and successfully integrating a portable wedge device could mark a significant breakthrough in preventive and rehabilitative care for musculoskeletal problems associated with the calf region. This innovative device can enhance the overall well-being and musculoskeletal health of individuals suffering from such issues, providing a more effective and convenient treatment solution.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients diagnosed with Trapezius tightness
* Age above 18-30
* Presence of active trigger points in the upper trapezius muscle
* Participants who are volunteer for the study
* Patients who suffer from shoulder pain and stiffness due to bad posture

Exclusion Criteria:

* History of whiplash injury
* History of head, neck, cervical spine or shoulder surgery
* History of cervical radiculopathy
* Diagnosed fibromyalgia and myopathy
* History of cancer
* Pregnancy Myofascial therapy within the past month
* Contraindication of dry needling and instrument-assisted soft tissue mobilization technique

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 12 Months
  A pain scale is a method used to quantify the level of discomfort a person is experiencing. It assesses a person's level of pain intensity on a scale from 0 to 10. The scale rates a person's level of discomfort at a particular moment and goes from '0', indicating no pain, to '10,' representing the worst pain imaginable. This simple yet efficient method is widely used to help healthcare professionals evaluate and treat pain.
Neck disability index (NDI) | 12 months
  To evaluate a patient's functional status, ten questions are asked about their condition, including pain, personal care, lifting, reading, headaches, focus, job, driving, sleeping, and recreation. Each category is scored from 0 to 5, where 0 indicates "No pain" and 5 indicates "Worst imaginable pain." The score can be multiplied by two to get a percentage score, with a maximum score of fifty.

CONTACTS AND LOCATIONS:
Locations (1):
- Faqraj Sharif Hospital (Trust) Physiotherapy and Orthopedic Department and Orian ABA Pakistan (Physiotherapy Department), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No